CLINICAL TRIAL: NCT00154089
Title: A Pilot Translational Study of Tetra-O-Methyl Nordihydroguaiaretic Acid (EM-1421) for the Treatment of Cervical Intraepithelial Neoplasia Induced by Human Papilloma Virus
Brief Title: A Pilot Study of EM-1421 for the Treatment of Cervical Intraepithelial Neoplasia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Erimos Pharmaceuticals (Industry)
Collaborators: University of Maryland, Baltimore County (Other); Planned Parenthood Delaware (Wilmington, DE) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EM-1421 #201
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2006-08

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: cervical intraepithelial neoplasia; CIN; HPV
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — terameprocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EM-1421 (Experimental): Administration of EM-1421 intravaginally once per week for 3 weeks
  Dose level of 45 mg/application (1% w/w) or 90 mg/application (2% w/w)
  Interventions: Drug: EM-1421

INTERVENTIONS:
Drug: EM-1421 — EM-1421 administered intravaginally every 3 weeks as 45 mg (1% w/w) EM-1421 or 90 mg (2% w/w) EM-1421
  Other Names: Terameprocol; M4N; Tetra-O-Methyl Nordihydroguaiaretic Acid

SUMMARY:
The primary objective of this study is to determine pilot safety and efficacy data for a topical formulation of EM-1421 applied to the cervix of patients with CIN 1, 2, or 3.

DETAILED DESCRIPTION:
This was an open-label, pilot Phase I/II dose evaluation and pharmacokinetic evaluation study to compare the safety and efficacy of terameprocol (45mg or 90mg/application)administered once per week for 3 weeks to the cervix uteri in patients with biopsy-proven CIN. Patients who met eligibility criteria visited the clinic weekly for terameprocol application. Patients kept a daily diary card record of genitourinary symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Negative pregnancy test
* Biopsy confirmed CIN 1, 2, or 3

Exclusion Criteria:

* Pregnancy or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-11; Primary Completion 2006-04 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Dept. of Family Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No